CLINICAL TRIAL: NCT01259895
Title: Effect os Sleep Restriction on Control of Food Intake and Metabolism of Obese Subjects
Brief Title: Effects of Time of Sleep Restriction in Obesity
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Collaborators: Associacao Fundo de Incentivo a Psicofarmcologia (Other); Centro de Estudos em Sonolência e Acidentes (Other)
Responsible Party: Principal Investigator, Iona Zalcman Zimberg, PhD student, Federal University of São Paulo
Other Study IDs: CEPE18; FAPESP2008/09565-2 (Other Grant/Funding Number: FAPESP)
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Obesity; Sleep Restriction; Appetite Regulation; Eating
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Obesity: BMI > 30kg/m2
- Normal weight: BMI between 19 and 24,9kg/m2

SUMMARY:
The purpose of this study is to determine the effect of different time of sleep restriction on control of food intake and metabolism of obese and normal subjects.

DETAILED DESCRIPTION:
The reduction of sleep time has now become a common habit, driven by the demands and opportunities of modern society. Some studies have suggested that sleep restriction would be an important factor in predisposing to obesity. However studies of sleep restriction in obese individuals have not yet been conducted. Still, the time of sleep restriction varies greatly between studies, making it difficult to compare results.

The investigators aim to recruit 20 young adults, 10 obese and 10 normal weight individuals. The study will be conducted as a randomized, crossover study with three conditions. Each participant will be subjected to reduction of the beginning of sleep (from 3-7h), reduction of the end of sleep (from 23-3h), and normal sleep (from 23-7h), in random order, for three consecutive nights.

In each condition, subjects will stay for 4 days in the laboratory. Three control meals will be offered. Visual analogue scales will be applied before and after each meal to assess hunger and appetite for different food categories. Blood samples will be collected hourly during 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* obese (BMI>30) and normal weight (BMI between 19 and 24,9)
* regular time of sleep between 6.5 and 8 hours

Exclusion Criteria:

* self-reported sleep problems (Pittsburgh Sleep Quality Index score >5);
* Obstructive sleep apnea (AHI > 5 in polysomnography)
* night work;
* variable sleep habits or habitual daytime naps;
* regular physical exercise (>3 hours/week);
* excessive intake of alcohol (>7 drinks/week);
* excessive intake of caffeine (>300 mg/day);
* smoking;
* substance abuse;
* use of prescription medications or over-the-counter drugs affecting sleep or metabolism;
* chronic diseases (e.g. cancer, asthma, back pain, thyroid disease, heart disease, diabetes, etc.)
* history of neurological, medical or sleep disorders;
* trans-meridian travelling the last month;
* chronotype: extreme morning or extreme evening
* unable to comply with the protocol.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: primary care clinic, community sample, residents of the city of Sao Paulo
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Appetite regulating hormones and stress hormones | Measured every hour over the course of 24 hours on day 3
  Hormones are sampled from blood

SECONDARY OUTCOMES:
Hunger and satiety | Measured every 4 hour over the course of 12 hours on day 2 and 3
  Hunger and saciety are measured using visual analogue scales before and after breakfast, lunch and dinner meal
Food intake | measured each meal
  The meal will be weighted before and after the breakfast, lunch and dinner. Energy and nutrient intake are assessed from the amount of the meal consumed.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tulio de Mello, PhD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Centro de Estudos em Psicobiologia e Exercicio (CEPE), São Paulo, São Paulo, Brazil